CLINICAL TRIAL: NCT02747004
Title: A Randomized, Open-Label, Phase 2 Study of Abemaciclib Plus Tamoxifen or Abemaciclib Alone, in Women With Previously Treated Hormone Receptor-Positive, HER2-Negative, Metastatic Breast Cancer
Brief Title: A Study of Abemaciclib (LY2835219) Plus Tamoxifen or Abemaciclib Alone in Women With Metastatic Breast Cancer
Acronym: Next MONARCH 1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16339; I3Y-MC-JPCG (Other: Eli Lilly and Company); 2016-000288-18 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abemaciclib + Tamoxifen (Experimental): Abemaciclib given orally every 12 hours (Q12H) in combination with tamoxifen given orally every day. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Tamoxifen
- Abemaciclib (Experimental): Abemaciclib given orally Q12H. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Abemaciclib + Prophylactic Loperamide (Experimental): Abemaciclib given orally Q12H in combination with prophylactic loperamide given orally. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Prophylactic Loperamide

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Tamoxifen — Administered orally
  Arms: Abemaciclib + Tamoxifen
Drug: Prophylactic Loperamide — Administered orally
  Arms: Abemaciclib + Prophylactic Loperamide

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of abemaciclib plus tamoxifen or abemaciclib alone in women with previously treated hormone receptor-positive (HR+), human epidermal growth factor receptor 2 negative (HER2-), metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HR+, HER2- breast cancer.
* Relapsed or progressed following endocrine therapy.
* Have received prior treatment with at least 2 chemotherapy regimens, of which at least 1 but no more than 2 have been administered in the metastatic setting.
* Have the presence of measureable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued previous therapies for cancer (including specifically, aromatase inhibitors, anti-estrogens, chemotherapy, radiotherapy, and immunotherapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (until the toxicity resolves to either baseline or at least Grade 1) except for residual alopecia or peripheral neuropathy.
* Have adequate organ function.
* Have negative serum pregnancy test within 7 days prior to the first dose of study treatment and agree to use highly effective precautions to prevent pregnancy during the study and for 3 weeks following last dose of study treatment.
* Are able to swallow oral medication.

Exclusion Criteria:

* Have clinical evidence or history of central nervous system metastasis.
* Have a personal history of any of the following conditions: syncope of either unexplained or cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
* Have active bacterial or fungal infection (that is, requiring intravenous antibiotics at the time of initiating study treatment) and/or detectable viral infection.
* Have received treatment with a prior cyclin-dependent kinase (CDK4) and CDK 6 inhibitor.
* Have a preexisting chronic condition resulting in persistent diarrhea.
* Have a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix or breast), unless in complete remission with no therapy for a minimum of 3 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (59):
- United States (5):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - University of Wisconsin Clinical Research Center, Madison, Wisconsin
- Argentina (6):
  - CENIT Centro de Neurociencias, Investigación y Tratamiento, CABA, Buenos Aires
  - Fundacion Ars Medica, San Salvador de Jujuy, Jujuy Province
  - Clinica Viedma, Viedma, Río Negro Province
  - Instituto de Oncología de Rosario, Rosario, Santa Fe Province
  - Centro Para la Atención Integral del Paciente Oncologico (CAIPO), San Miguel de Tucumán, Tucumán Province
  - Sanatorio Parque, Salta
- Austria (3):
  - Medizinische Universitaet Graz, Graz, Styria
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
  - AKH, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - VITAZ, Sint-Niklaas, Oost-Vlaanderen
  - Grand Hopital de Charleroi-Site Notre-Dame, Charleroi
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- Brazil (4):
  - Hospital São Lucas - PUCRS - ONCOLOGY, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Clinica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária LTDA, São Paulo
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno, Czech Republic
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Fakultni Poliklinika VFN, Prague
  - Fakultni Nemocnice v Motole, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- France (2):
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
- Germany (2):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Kath. Marienkrankenhaus gGmbH, Hamburg
- Italy (4):
  - Polic.Umberto I -Univ. La Sapienza, Roma, Rome
  - Ospedale Sacro Cuore Don G. Calabria, Negrar, Verona
  - Ospedale Bellaria - Azienda USL di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
- Mexico (4):
  - Neurociencias Estudios Clinicos, Culiacán, Sinaloa
  - Centro Hemato Oncologico Privado, San Bernardino, Toluca
  - Grupo Medico Camino Sc, Mexico City
  - Oaxaca Site Management Organization, Oaxaca City
- Russia (3):
  - Republic Oncology Dispensary of MoH of Republic Tatarstan, Kazan'
  - St-Petersburg scientifical practical center of specialized medical care, Saint Petersburg
  - Saint-Petersburg city clinical oncology dispensary, Saint Petersburg
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Clinic I Provincial, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (5):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- Turkey (Türkiye) (5):
  - Erciyes University Faculty of Medicine, Kayseri, Melikgazi
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Hacettepe University Faculty of Medicine, Ankara
  - Medipol Mega University Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Hamilton E, Cortes J, Ozyilkan O, Chen SC, Petrakova K, Manikhas A, Jerusalem G, Hegg R, Huober J, Zhang W, Chen Y, Martin M. nextMONARCH Phase 2 randomized clinical trial: overall survival analysis of abemaciclib monotherapy or in combination with tamoxifen in patients with endocrine-refractory HR + , HER2- metastatic breast cancer. Breast Cancer Res Treat. 2022 Aug;195(1):55-64. doi: 10.1007/s10549-022-06662-9. Epub 2022 Jul 12. PMID 35829935
- See also: A Study of Abemaciclib (LY2835219) Plus Tamoxifen or Abemaciclib Alone in Women With Metastatic Breast Cancer (nextMONARCH 1) — https://trials.lillytrialguide.com/en-US/trial/11MY3TKjOeIWgmIkemWkyM

RESULTS

PARTICIPANT FLOW:
Groups:
- 150mg Abemaciclib + 20mg Tamoxifen: Participants received oral dose of 150 milligrams (mg) Abemaciclib every 12 hours (Q12H) along with 20mg Tamoxifen every 24 hours (QD) on days 1 to days 28 of a 28 day cycle.
- 150mg Abemaciclib: Participants received oral dose of 150 milligrams (mg) Abemaciclib every 12 hours (Q12H) on days 1 to days 28 of a 28 day cycle.
- 200mg Abemaciclib + 2mg Prophylactic Loperamide: Participants received oral dose of 200 milligrams (mg) Abemaciclib every 12 hours (Q12H) along with 2mg Prophylactic Loperamide on days 1 to days 28 of a 28 day cycle.
  Note: During Cycle 1, 2mg prophylactic loperamide was administered orally with the first dose of abemaciclib daily. During Cycle 2 and beyond, loperamide was administered at investigator's discretion and/or if clinically indicated.
Period: Overall Study
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Started | 78 | 79 | 77
Received at Least One Dose of Study Drug | 78 | 79 | 77
Completed | 21 | 30 | 30
Not Completed | 57 | 49 | 47
Not completed — Withdrawal by Subject | 8 | 5 | 4
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — on study treatment/follow-up | 48 | 42 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide | Total
Number analyzed (Participants) | 78 | 79 | 77 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.28 (12.47) | 56.18 (12.24) | 55.86 (11.03) | 55.44 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 79 | 77 | 234
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 20 | 21 | 57
  Not Hispanic or Latino | 55 | 45 | 46 | 146
  Unknown or Not Reported | 7 | 14 | 10 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 4 | 11
  Asian | 8 | 6 | 10 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 63 | 64 | 60 | 187
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival time was measured from the date of randomization to the date of investigator-determined objective progression as defined by RECIST v1.1, or death from any cause, whichever occurred first. Progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Participants who have neither progressed nor died were censored at the day of their last radiographic tumor assessment (if available) or date of randomization if no post baseline radiographic assessment is available.
Time Frame: Baseline to Objective Disease Progression or Death from Any Cause (Up to 21 Months)
Population: All randomized participants who received at least one dose of study drug. Censored participants: 21 in Abemaciclib 150 mg + Tamoxifen 20mg; 25 in Abemaciclib 150 mg; 22 in Abemaciclib 200mg.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- 200mg Abemaciclib + 2mg Prophylactic Loperamide: Participants received oral dose of 150 milligrams (mg) Abemaciclib every 12 hours (Q12H) along with 2mg Prophylactic Loperamide on days 1 to days 28 of a 28 day cycle.
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 78 | 79 | 77
Months | 9.07 [6.90 to 10.95] | 6.48 [4.77 to 9.21] | 7.43 [5.42 to 9.17]
Statistical Analysis 1: Comparison: 150mg Abemaciclib + 20mg Tamoxifen vs 200mg Abemaciclib + 2mg Prophylactic Loperamide; Test type: Superiority; p = 0.2930, Log Rank — Two-sided P-value; Stratified by the randomization factors of presence of liver metastases and prior use of Tamoxifen in the advanced/metastatic setting
Statistical Analysis 2: Comparison: 150mg Abemaciclib vs 200mg Abemaciclib + 2mg Prophylactic Loperamide; Test type: Other — Informal phase 2 non-inferiority; Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.045, 95% CI 2-sided [0.711 to 1.535]

2. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: Objective response rate was defined as the percentage of participants with CR or PR according to RECIST v1.1. CR was defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the LD (longest diameter) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression (Up to 21 Months)
Population: All randomized participants who received at least one dose of study drug and had PR/CR data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 78 | 79 | 77
Percentage of participants | 34.6 [24.1 to 45.2] | 24.1 [14.6 to 33.5] | 32.5 [22 to 42.9]

3. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date of first evidence of a CR or PR to the date of objective progression or death from any cause, whichever is earlier as defined by Recist v1.1. CR was defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up to 21 Months)
Population: All randomized participants who received at least one dose of study drug and achieved CR or PR.
  Censored participants: 9 in Abemaciclib 150 mg + Tamoxifen 20mg; 9 in Abemaciclib 150 mg; 11 in Abemaciclib 200mg.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 27 | 19 | 25
Months | 7.40 [3.88 to 9.27] | 9.21 [3.72 to NA] — Upper bound not estimable. | 7.46 [5.56 to 10.92]

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Baseline to Death from Any Cause (Approximately 36 Months)
Reporting Status: Not Posted

5. Secondary Outcome: Pharmacokinetics (PK): Mean Single Dose Concentration of Abemaciclib and Its Metabolites
Description: Mean single dose concentrations of Abemaciclib and its metabolites (M2 & M20) are reported.
Time Frame: Cycle (C) 1 Day (D) 1 post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Millilitre (ng/mL)
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 19 | 13 | 20
Nanogram per Millilitre (ng/mL)
  Abemaciclib (C1D1): number analyzed (Participants) | 17 | 10 | 15
  Abemaciclib (C1D1) | 10.9 (231) | 3.05 (95.4) | 8.59 (440)
  M2 (C1D1): number analyzed (Participants) | 18 | 9 | 13
  M2 (C1D1) | 6.05 (123) | 2.14 (60.1) | 6.85 (237)
  M20 (C1D1) | 6.50 (132) | 2.54 (54.5) | 7.91 (220)

6. Secondary Outcome: Pharmacokinetics (PK): Steady State Concentration of Abemaciclib and Its Metabolites
Description: Mean steady state concentrations of Abemaciclib and its metabolites (M2 & M20) are reported.
  C=Cycle D= Day
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1 post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Millilitre (ng/mL)
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 55 | 56 | 46
Nanogram per Millilitre (ng/mL)
  Abemaciclib (C1D15) | 214 (66.4) | 256 (58.8) | 314 (74.3)
  M2 (C1D15) | 96.5 (53.9) | 108 (45.6) | 147 (47.1)
  M20 (C1D15) | 180 (51.1) | 199 (41.0) | 251 (48.5)
  Abemaciclib (C2D1): number analyzed (Participants) | 55 | 48 | 30
  Abemaciclib (C2D1) | 98.9 (196) | 182 (129) | 220 (154)
  M2 (C2D1): number analyzed (Participants) | 54 | 48 | 30
  M2 (C2D1) | 56.1 (88.0) | 85.4 (62.1) | 105 (98.5)
  M20 (C2D1): number analyzed (Participants) | 55 | 48 | 29
  M20 (C2D1) | 100 (103) | 149 (78.9) | 164 (171)
  Abemaciclib (C2D15): number analyzed (Participants) | 49 | 39 | 27
  Abemaciclib (C2D15) | 135 (115) | 157 (173) | 175 (136)
  M2 (C2D15): number analyzed (Participants) | 48 | 39 | 27
  M2 (C2D15) | 62.3 (79.0) | 71.7 (97.9) | 95.4 (73.9)
  M20 (C2D15): number analyzed (Participants) | 48 | 39 | 27
  M20 (C2D15) | 120 (76.2) | 128 (121) | 154 (101)
  Abemaciclib (C3D1): number analyzed (Participants) | 43 | 32 | 22
  Abemaciclib (C3D1) | 125 (64.3) | 177 (42.0) | 207 (49)
  M2 (C3D1): number analyzed (Participants) | 43 | 32 | 22
  M2 (C3D1) | 60.6 (39.6) | 78.4 (38.2) | 95.8 (44.2)
  M20 (C3D1): number analyzed (Participants) | 43 | 32 | 22
  M20 (C3D1) | 109 (39.4) | 146 (37.7) | 171 (36.6)

7. Secondary Outcome: PK: Mean Single Dose Concentration of Tamoxifen and Endoxifen
Description: Mean single dose concentrations of Tamoxifen and its metabolite (Endoxifen) were reported.
Time Frame: Cycle 1 Day 1 post dose
Population: All randomized participants who received at least one dose of study drug along with Tamoxifen and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen
Number analyzed (Participants) | 21
ng/mL
  Tamoxifen (C1D1) | 7.47 (116)
  Endoxifen (C1D1): number analyzed (Participants) | 2
  Endoxifen (C1D1) | NA (NA) — Geometric Mean was not able to be calculated due to small sample size (2 Participants). Individual values = 0.653 ng/mL, 3.8 ng/mL.

8. Secondary Outcome: PK: Multiple Dose Concentration of Tamoxifen and Endoxifen
Description: Mean multiple dose concentrations of Tamoxifen and its metabolite (Endoxifen) were reported.
Time Frame: Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1 post dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen
Number analyzed (Participants) | 48
ng/mL
  Tamoxifen (C1D15) | 84.5 (41.6)
  Endoxifen (C1D15) | 4.76 (99.7)
  Tamoxifen (C2D1): number analyzed (Participants) | 45
  Tamoxifen (C2D1) | 98.7 (50.2)
  Endoxifen (C2D1): number analyzed (Participants) | 45
  Endoxifen (C2D1) | 7.41 (89.5)
  Tamoxifen (C2D15): number analyzed (Participants) | 44
  Tamoxifen (C2D15) | 109 (51.9)
  Endoxifen (C2D15): number analyzed (Participants) | 44
  Endoxifen (C2D15) | 9.17 (73.7)
  Tamoxifen (C3D1): number analyzed (Participants) | 34
  Tamoxifen (C3D1) | 112 (60.2)
  Endoxifen (C3D1): number analyzed (Participants) | 34
  Endoxifen (C3D1) | 10.3 (84.8)

9. Secondary Outcome: Change From Baseline in Symptom Burden on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 self-reported general cancer instrument consists of 30 items covered by 1 of 3 dimensions:
  1. Global health status/quality of life (2 items) with scores ranging from 1 (Very Poor) to 7 (Excellent).
  2. Functional scales (15 total items addressing either physical, role, emotional, cognitive, or social functioning), each item scores ranging from 1 (not at all) to 4 (very much)
  3. Symptom scales (13 total items addressing either fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, or financial impact), each item scores ranging from 1 (not at all) to 4 (very much).
  Raw scores are linearly converted to a 0-100 scale with higher scores reflecting higher levels of function/QOL or higher levels of symptom burden.
Time Frame: Baseline, 21 Months
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-C30 score.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 77 | 75 | 76
score on a scale
  Global Health Status: number analyzed (Participants) | 76 | 75 | 76
  Global Health Status | 1.56 (1.83) | 4.56 (1.90) | -2.77 (1.91)
  Functional Scales (Physical Functioning) | -2.01 (1.59) | -1.05 (1.68) | -2.65 (1.68)
  Functional Scales (Role Functioning) | -0.44 (2.18) | -3.95 (2.30) | -5.87 (2.29)
  Functional Scales (Emotional Functioning): number analyzed (Participants) | 76 | 75 | 76
  Functional Scales (Emotional Functioning) | 4.40 (1.88) | 2.58 (1.95) | 1.86 (1.95)
  Functional Scale (Cognitive Functioning): number analyzed (Participants) | 76 | 75 | 76
  Functional Scale (Cognitive Functioning) | 0.14 (1.37) | -1.31 (1.44) | -2.39 (1.43)
  Functional Scales (Social Functioning): number analyzed (Participants) | 76 | 75 | 76
  Functional Scales (Social Functioning) | 3.23 (2.08) | -0.53 (2.16) | -0.94 (2.16)
  Symptom Scales (Fatigue) | 2.39 (2.05) | 2.77 (2.15) | 4.0 (2.16)
  Symptom Scales (Nausea and Vomiting) | 5.59 (1.63) | 5.30 (1.73) | 5.09 (1.71)
  Symptom Scales (Pain): number analyzed (Participants) | 76 | 75 | 76
  Symptom Scales (Pain) | -3.09 (2.20) | -1.43 (2.30) | -2.01 (2.29)
  Symptom Scales (Dyspnoea) | 4.21 (1.79) | -3.49 (1.89) | -2.0 (1.87)
  Symptom Scales (Insomnia) | -5.02 (2.21) | -3.43 (2.36) | -2.98 (2.35)
  Symptom Scales (Appetite Loss) | 5.82 (2.38) | 1.87 (2.50) | 7.76 (2.50)
  Symptom Scales (Constipation): number analyzed (Participants) | 76 | 74 | 76
  Symptom Scales (Constipation) | -0.28 (1.57) | -6.29 (1.71) | 0.08 (1.67)
  Symptom Scales (Diarrhoea): number analyzed (Participants) | 76 | 75 | 76
  Symptom Scales (Diarrhoea) | 13.31 (1.97) | 20.17 (2.10) | 17.43 (2.09)
  Symptom Scales (Functional Difficulties): number analyzed (Participants) | 76 | 75 | 76
  Symptom Scales (Functional Difficulties) | -7.56 (2.00) | -3.81 (2.08) | -0.09 (2.07)

10. Secondary Outcome: Change From Baseline in Pain and Symptom Burden Assessment on the Modified Brief Pain Inventory-Short Form (mBPI-sf)
Description: mBPI-sf is an 11-item instrument used as a multiple-item measure of cancer pain intensity. In addition to pain intensity (4 items), the mBPI-sf is designed for participants to record the presence of pain in general, pain relief, and pain interference with function (general activity, mood, ability to walk, ability to perform normal work, relations with others, sleep, enjoyment of life). Responses for the mBPI-sf items are captured through the use of 11-point numeric rating scales anchored at 0 (no pain or does not interfere) and 10 (pain as bad as you can imagine or completely interferes). The mBPI-sf recall period is 24 hours and typical completion time for this instrument is less than 5 minutes.
Time Frame: Baseline, 21 Months
Population: All randomized participants who received at least one dose of study drug and had baselines and post baseline mBPI-sf measurement.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
Number analyzed (Participants) | 78 | 76 | 75
score on a scale
  Pain at its Worst in Last 24 Hours | -0.53 (0.20) | -0.43 (0.21) | -0.43 (0.21)
  Pain at its Least in Last 24 Hours | -0.09 (0.15) | -0.01 (0.16) | 0.14 (0.16)
  Pain on the Average: number analyzed (Participants) | 78 | 75 | 75
  Pain on the Average | -0.34 (0.16) | -0.20 (0.17) | -0.11 (0.17)
  Pain Right Now | -0.28 (0.17) | -0.18 (0.17) | -0.04 (0.17)
  Mean Interference Score: number analyzed (Participants) | 77 | 76 | 75
  Mean Interference Score | -0.09 (0.18) | 0.03 (0.18) | 0.16 (0.18)

ADVERSE EVENTS:
Time Frame: Up to 21 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 150mg Abemaciclib + 20mg Tamoxifen | 150mg Abemaciclib | 200mg Abemaciclib + 2mg Prophylactic Loperamide
All-Cause Mortality (participants affected / at risk) | 18/78 | 28/79 | 29/77
Serious Adverse Events (participants affected / at risk) | 16/78 | 16/79 | 21/77
Other Adverse Events (participants affected / at risk) | 73/78 | 77/79 | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150mg Abemaciclib + 20mg Tamoxifen (N=78) | 150mg Abemaciclib (N=79) | 200mg Abemaciclib + 2mg Prophylactic Loperamide (N=77)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150mg Abemaciclib + 20mg Tamoxifen (N=78) | 150mg Abemaciclib (N=79) | 200mg Abemaciclib + 2mg Prophylactic Loperamide (N=77)
Anaemia (Blood and lymphatic system disorders) | 30 (63) | 24 (36) | 31 (68)
Leukopenia (Blood and lymphatic system disorders) | 9 (24) | 10 (23) | 6 (9)
Neutropenia (Blood and lymphatic system disorders) | 21 (64) | 20 (46) | 18 (51)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (18) | 1 (1) | 5 (5)
Dry eye (Eye disorders) | 0 (0) | 4 (4) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 6 (7) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 16 (21) | 11 (17) | 19 (21)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 8 (10) | 6 (7)
Constipation (Gastrointestinal disorders) | 10 (16) | 9 (13) | 25 (28)
Diarrhoea (Gastrointestinal disorders) | 41 (161) | 53 (244) | 47 (140)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 3 (3) | 4 (6)
Flatulence (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 24 (48) | 26 (47) | 33 (50)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 4 (7) | 4 (6)
Toothache (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (34) | 20 (62) | 20 (34)
Asthenia (General disorders) | 14 (26) | 14 (20) | 6 (7)
Fatigue (General disorders) | 22 (32) | 17 (30) | 21 (41)
Mucosal inflammation (General disorders) | 5 (8) | 3 (4) | 2 (2)
Oedema peripheral (General disorders) | 3 (4) | 6 (8) | 7 (7)
Pyrexia (General disorders) | 7 (8) | 5 (7) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 4 (6) | 4 (5)
Urinary tract infection (Infections and infestations) | 7 (8) | 5 (6) | 5 (5)
Alanine aminotransferase increased (Investigations) | 6 (10) | 4 (6) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 8 (12) | 4 (5) | 7 (8)
Blood alkaline phosphatase increased (Investigations) | 4 (10) | 3 (4) | 4 (4)
Blood creatinine increased (Investigations) | 14 (35) | 7 (15) | 8 (11)
Gamma-glutamyltransferase increased (Investigations) | 3 (5) | 5 (13) | 3 (7)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (20) | 3 (4)
Neutrophil count decreased (Investigations) | 11 (22) | 21 (71) | 22 (81)
Platelet count decreased (Investigations) | 8 (14) | 9 (22) | 22 (49)
Weight decreased (Investigations) | 5 (9) | 9 (10) | 5 (6)
White blood cell count decreased (Investigations) | 12 (26) | 18 (56) | 15 (52)
Decreased appetite (Metabolism and nutrition disorders) | 20 (29) | 12 (21) | 17 (27)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 (22) | 3 (3) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (9) | 3 (3) | 6 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 8 (11) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (7) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 11 (14) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (8) | 7 (12) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 5 (7) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (5) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 7 (11) | 6 (7) | 7 (7)
Paraesthesia (Nervous system disorders) | 3 (5) | 4 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7) | 10 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 12 (15) | 5 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (9) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7) | 4 (4)
Hot flush (Vascular disorders) | 6 (9) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT02747004/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT02747004/SAP_001.pdf